CLINICAL TRIAL: NCT05180201
Title: Safety, Tolerability and Effects on the Microbiome of Neonatal Administration of Lactiplantibacillus Plantarum ATCC 202195 With or Without Fructooligosaccharide for One or Seven Days: a Phase II Randomized Placebo-controlled Trial in Dhaka, Bangladesh
Brief Title: SEPSIS: L. Plantarum Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Child Health Research Foundation, Bangladesh (Other); Boston University (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Daniel Roth, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1000072200
Record Dates: First submitted 2021-11-25; First posted 2022-01-06 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Microbial Colonization; Tolerance; Safety Issues; Infant ALL
Keywords: Probiotic; Synbiotic; Young infants; Bangladesh
MeSH Terms: conditions — Communicable Diseases | interventions — Synbiotics; Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, parallel-design multi-arm trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation concealment and blinding of participants, study personnel, and investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- LP7+FOS (Experimental): Once daily oral administration of L. plantarum ATCC 202195 (10^9 CFU/day) with 150mg fructooligosaccharide (FOS) and 100mg maltodextrin, for 7 days.
  Interventions: Dietary Supplement: Synbiotic
- LP7 (Experimental): Once daily oral administration of L. plantarum ATCC 202195 (10^9 CFU/day) plus 250mg maltodextrin, for 7 days.
  Interventions: Dietary Supplement: Probiotic
- LP1+FOS (Experimental): Once daily oral administration of L. plantarum ATCC 202195 (10^9 CFU/day) with 150mg FOS and 100mg maltodextrin, for one day, followed by 6 days of placebo (250mg maltodextrin).
  Interventions: Dietary Supplement: Synbiotic; Other: Placebo
- LP1 (Experimental): Once daily oral administration of L. plantarum ATCC 202195 (10^9 CFU/day) plus 250mg maltodextrin for one day, followed by 6 days of placebo (250 mg maltodextrin).
  Interventions: Dietary Supplement: Probiotic; Other: Placebo
- Placebo (Placebo Comparator): Once daily oral administration of placebo (250 mg maltodextrin), for 7 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic — Lactiplantibacillus plantarum ATCC 202195 with fructooligosaccharide
  Arms: LP1+FOS; LP7+FOS
Dietary Supplement: Probiotic — Lactiplantibacillus plantarum ATCC 202195
  Arms: LP1; LP7
Other: Placebo — Maltodextrin
  Arms: LP1; LP1+FOS; Placebo

SUMMARY:
Sepsis is a life-threatening clinical syndrome and a leading cause of neonatal deaths worldwide. The burden of neonatal sepsis and severe infection (SI) is particularly high in areas of South Asia and other resource-limited settings. The goal of the Synbiotics for the Early Prevention of Severe Infections in Infants (SEPSIS) phase II L. plantarum trial is to generate knowledge on the safety, tolerability and effects on the microbiome of Lactiplantibacillus plantarum, with or without fructooligosaccharide, in infants (birth to 60 days of age) in Dhaka, Bangladesh. All data generated will support the design and implementation of a phase III trial to test the efficacy of the probiotic/synbiotic or other interventions for the prevention of SI, promotion of optimal growth and development, and effects on other health outcomes in early infancy.

DETAILED DESCRIPTION:
As a leading cause of neonatal morbidity and mortality, sepsis poses a common and serious threat for neonates. In 2017, sepsis, meningitis, and pneumonia accounted for an estimated 540,000 newborn deaths worldwide, or approximately one-fifth of the world's annual neonatal deaths. Previous studies have suggested that South Asia has a relatively high incidence of possible serious bacterial infection (pSBI) in young infants, particularly in areas where neonatal and under-five mortality rates are highest.

Recent randomized controlled trials (RCTs), including the Panigrahi et al. community-based trial in India, have demonstrated beneficial effects of probiotics and/or prebiotics, compared to placebo, for preventing infections in preterm and/or LBW infants. This is particularly important in low- and middle-income countries in Africa and South Asia, where low-cost preventative interventions to reduce the burden of SI (e.g., probiotics or synbiotics) could have an important impact on the burden of morbidity and mortality in young infants. However, there are limited data regarding the safety, tolerability and efficacy of L. plantarum ATCC 202195 in the general population of infants (rather than selected groups of preterm or hospitalized newborns) in South Asia.

This phase II trial will generate new evidence about the safety, tolerability and colonization effects of L. plantarum ATCC 2020195 in young infants (birth to 60 days of age) in Dhaka, Bangladesh. The aims of this study are to:

1. Estimate the effect of neonatal oral administration of Lactiplantibacillus plantarum (L. plantarum) ATCC 202195 (10^9 CFU/day) with or without fructooligosaccharide (FOS), versus placebo, on the absolute and relative stool abundance of L. plantarum ATCC 202195 from 14 to 60 days of age. Primary analyses will examine the effect of a 7-day regimen of L. plantarum ATCC 202195 with FOS (LP7+FOS), and secondary analyses will examine a 7-day regimen of L. plantarum ATCC 202195 without FOS (LP7), a 1-day regimen of L. plantarum ATCC 202195 with FOS (LP1+FOS), or a 1-day regimen of L. plantarum ATCC 202195 without FOS (LP1).
2. Determine if the absolute and relative stool abundance of L. plantarum ATCC 202195 from 14 to 60 days of age in Bangladeshi infants following LP1+FOS is not lower than the abundance achieved with LP7+FOS. Secondary analyses will assess the non-inferiority of the 1- and 7-day LP regimens without FOS (LP1 or LP7, respectively) compared to LP7+FOS.
3. Describe and compare the incidence and patterns of sustained and transient L. plantarum ATCC 202195 colonization (based on absolute and relative stool abundance) up to 6 months of age following administration of LP7+FOS, LP7, LP1+FOS or LP1, versus placebo, in Bangladeshi infants.
4. Assess the safety of LP7+FOS, LP7, LP1+FOS or LP1, versus placebo, during the first 60 days of age based on a) incidence of severe infection (SI) episodes associated with Lactobacillus spp.; b) incidence of detectable L. plantarum ATCC 202195 DNA in blood; c) adverse alterations in one or more biochemical or hematological parameters; and d) clinical serious adverse events.
5. Estimate the effects of LP7+FOS, LP7, LP1+FOS or LP1, versus placebo, on stool pH and concentrations of stool inflammatory markers during the first 60 days of life.
6. Assess the tolerability of LP7+FOS, LP7, LP1+FOS or LP1, versus placebo, following ingestion of the investigational product and during the period of administration (up to 21 days of age), based on frequencies and/or durations of crying time, fussiness, abdominal distention, vomiting and diarrhea.
7. Evaluate the effect of LP7+FOS, LP7, LP1+FOS or LP1, versus placebo, on stool iron content and antioxidant capacity (14 days of age) and iron status in infants (60 days of age).
8. Estimate effects of LP7+FOS, LP7, LP1+FOS and LP1, versus placebo, on infant linear growth, ponderal growth and head circumference up to 6 months of age.
9. Explore the effects of LP7+FOS, LP7, LP1+FOS or LP1, versus placebo, on the microbial community structure and diversity and metabolome of the infant's microbiota during the first 60 days of life and at 3 and 6 months of life.
10. Compare the absolute and relative stool abundance of L. plantarum ATCC 202195 in mothers and siblings of infants administered LP7+FOS, LP7, LP1+FOS, LP1, versus placebo, up to 60 days of age in the infant.
11. Assess the possible modes of cross-contamination by L. plantarum ATCC 202195 in two public hospitals, field offices, laboratories and in households within the trial catchment area in Dhaka, Bangladesh.

Study personnel will conduct active and passive clinical surveillance and routine specimen collection (e.g. stool, nasal, blood etc.). Additional specimen collection may also be triggered in the event of physician-confirmed clinical severe infection, or if infants meet the case definition of LRTI (fast breathing with at least one of the following: cough, nasal congestion, or runny nose) or are hospitalized with diarrhea and/or vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Infants up to and including four days of age*
* Infant delivered at a study hospital
* Orally feeding currently**
* Informed consent by parent or guardian
* Intends to maintain residence within the defined catchment areas (upon discharge from hospital) until 60 days of age.

Exclusion Criteria:

* Birthweight < 1500 grams***
* Death or major surgery considered to be highly probable within first week of life****
* Major congenital anomaly of the gastrointestinal tract
* Maternal HIV infection and/or history of mother ever receiving anti-retroviral drug(s) for presumed HIV infection*****
* Current mechanical ventilation and/or cardiac support (e.g., inotropes) and/or administration/prescription of parenteral antibiotics*
* Any prenatal or postpartum use of non-dietary probiotic supplement by mother during current pregnancy******
* Any postnatal administration of non-dietary probiotic or prebiotic supplements to infant
* Current participation of the infant in another clinical trial
* Resides in the same household as another infant previously enrolled in the study, or any study within the research platform, who is currently <60 days of age; however, twins may all be enrolled simultaneously in this trial.
* Multiple gestation for which the number of liveborn infants from the same pregnancy exceeds two (i.e., triplets or higher order multiples).

'*Day of birth is considered day 0 of life. Therefore, the infant could be enrolled on days 0, 1, 2, 3 or 4 of life.

'**These criteria are time-varying, so will be reassessed on a daily basis until no longer eligible for another reason (i.e., beyond day 4 of life) as long as the infant remains potentially eligible by other criteria. Orally feeding is defined as being able to take a probiotic or synbiotic supplement by mouth on a daily basis.

'***Current infant weight, as measured and documented by study personnel, will be used if birth weight is missing, illegibly recorded, or suspected of being an error (e.g., implausible value, discrepancy of greater than 15% between documented birth weight and measured screening weight).

'**** Major surgery as an operative procedure to explore and/or repair an organ or tissue that is performed under general anaesthesia. Examples relevant to the neonatal period include: ligation of patent ductus arteriosus, repair of abdominal wall defects, repair bowel perforation due to of necrotizing enterocolitis, repair of tracheoesophageal fistula and/or esophageal atresia, and repair of myelomeningocele. Conversely, examples of common procedures in newborns not considered major surgery include circumcision, tongue tie release, removal of extra digit (polydactyly).

'*****Although HIV in very young infants will be rare in this context, there is a low but non-zero theoretical risk that a baby born to an HIV positive mother could be significantly compromised, particularly in cases where in utero transmission occurred earlier in pregnancy. Both the HIV positive mother and infant are expected to represent a unique population in regards to their respective microbiomes, and excluding them should not affect generalizability of results to the population as a whole. The number of HIV positive infants is anticipated to be too low to conduct sub-group analyses and thus, it would not be possible to make meaningful inferences about this population, even if they were to be included in the study. Testing for HIV infection will not be performed as a study procedure; therefore, this criterion will be based on information available from the medical record.

'******Non-dietary probiotic supplement is a commercial (store-bought) probiotic product that is consumed in the form of a capsule, powder, liquid, etc., although it may be mixed into a food or drink at the time of consumption. In contrast, a dietary probiotic is an ingredient of a food or beverage that either occurs naturally or is added during home production or the commercial manufacturing process (e.g., yoghurt or fermented drinks).

Ages: 0 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 519 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Average absolute abundance of L. plantarum ATCC 202195 in stool, measured as cells/g faces or cells/ng DNA | Up to 60 days of age
  Absolute abundance (AA) of L. plantarum ATCC 202195 (LP202195) in stool samples refers to the log number of cells of LP202195 per mass of total extracted DNA and/or mass of stool as measured by qPCR. AA will be defined as the stool abundance of LP202195 from day 14 to 60 of age, based on up to 5 post-intervention period stool samples. However, additional analyses will involve variations on the outcome definition based on a) the age at which samples were collected and, b) timing of collection in relation to the intervention period.
Average relative abundance of L. plantarum ATCC 202195 in stool, measured as a ratio | Up to 60 days of age
  Relative abundance (RA) refers to the proportion of LP202195 relative to the total bacterial load, where total bacterial load is determined by the absolute quantification of 16S rRNA gene copies as measured by qPCR. RA will be defined as the stool abundance of LP202195 from day 14 to 60 of age, based on up to 5 post-intervention period stool samples. However, additional analyses will involve variations on the outcome definition based on a) the age at which samples were collected and, b) timing of collection in relation to the intervention period.
Other microbial efficacy outcomes: L. plantarum ATCC 202195 Colonization | Up to 60 days of age
  Colonization is a dichotomous variable (colonized or not) defined as a stool AA of L. plantarum ATCC 202195 that exceeds a specified threshold. Empirical distributions across all groups will be used to derive plausible thresholds of colonization based on qPCR.
Other microbial efficacy outcomes: Time to L. plantarum ATCC 202195 colonization | Up to 60 days of age
  Time to colonization is defined as the earliest age (in days) at which an infant's stool had an AA value that exceeded the threshold for colonization based on qPCR.
Other microbial efficacy outcomes: Stool inflammatory markers | Up to 60 days of age
  Stool inflammatory markers include stool concentrations of calprotectin (µg/g) and myeloperoxidase (ng/ml) derived from standard curves based on ELISAs.
Other microbial efficacy outcomes: Stool pH | Up to 60 days of age
  Stool pH will be expressed as a continuous outcome and categorized as low if stool pH <4.5.

SECONDARY OUTCOMES:
Cumulative incidence of episodes of culture-confirmed lactobacillus spp. related severe infection (Primary clinical safety outcome) | Up to 60 days of age
  An episode of severe infection (SI) for which the presumptive cause is Lactobacilli, implying isolation of lactobacillus spp. in blood (bacteremia), CSF (meningitis) or urine (urinary tract infection) based on conventional microbiological culture.
Cumulative incidence of episodes of detectable L. plantarum ATCC 202195 bacteremia (ancillary safety measure, IF FEASIBLE) | Up to 60 days of age
  Presence of detectable L. plantarum ATCC 202915 in blood using ddPCR.
Frequency of hemoglobin (g/L or g/dL) below reference limit | Up to 60 days of age
  Hemoglobin will be measured in routinely collected samples, and the proportion of values above the reference limit will be compared across intervention groups.
Frequency of white blood cell count (10^9 cells/L) above or below reference limit | Up to 60 days of age
  White blood cell count will be measured in routinely collected samples, and the proportion of values above the reference limit will be compared across intervention groups.
Frequency of platelet count (10^9 cells/L) above or below reference limit | Up to 60 days of age
  Platelet count will be measured in routinely collected samples, and the proportion of values above the reference limit will be compared across intervention groups.
Average hemoglobin (g/L or g/dL) | Up to 60 days of age
  Hemoglobin will be measured in routinely collected samples, and the averages will be compared across intervention groups.
Average white blood cell count (10^9 cells/L) | Up to 60 days of age
  White blood cell count will be measured in routinely collected samples, and the averages will be compared across intervention groups.
Average platelet count (10^9 cells/L) | Up to 60 days of age
  Platelet cell count will be measured in routinely collected samples, and the averages will be compared across intervention groups.
Frequency of serum C-reactive protein (mg/L) above reference limit | Up to 60 days of age
  C-reactive protein will be measured in routinely collected samples, and the proportion of values above the reference limit will be compared across intervention groups.
Average concentration of serum C-reactive protein (mg/L) | Up to 60 days of age
  C-reactive protein will be measured in routinely collected samples, and group-average concentrations will be compared across intervention groups.
Frequency of serum procalcitonin (ug/L) above reference limit | Up to 60 days of age
  Procalcitonin will be measured in routinely collected samples, and the proportion of values above the reference limit will be compared across intervention groups.
Average concentration of serum procalcitonin (ug/L) | Up to 60 days of age
  Procalcitonin will be measured in routinely collected samples, and group-average concentrations will be compared across intervention groups.
Average concentration of serum creatinine (μmol/L) | Up to 60 days of age
  Creatinine will be measured in routinely collected samples, and group-average concentrations will be compared across intervention groups.
Average concentration of serum Alanine Aminotransferase (ALT) (U/L) | Up to 60 days of age
  ALT will be measured in routinely collected samples, and group-average concentrations will be compared across intervention groups.
Average concentration of serum total bilirubin (μmol/L) | Up to 60 days of age
  Bilirubin will be measured in routinely collected samples, and group-average concentrations will be compared across intervention groups.
Average concentration of serum conjugated bilirubin (μmol/L) | Up to 60 days of age
  Bilirubin will be measured in routinely collected samples, and group-average concentrations will be compared across intervention groups.
Average concentration of serum albumin (g/L) | Up to 60 days of age
  Albumin will be measured in routinely collected samples, and group-average concentrations will be compared across intervention groups.
Average concentration of glucose (mmol/L) | Up to 60 days of age
  Glucose will be measured in routinely collected samples, and group-average concentrations will be compared across intervention groups.
Safety outcomes: Serious adverse events | Up to 60 days of age
  Serious adverse events (SAE) will be compared between groups for infants during the first 60 days of life.
Frequency of dripping/drooling or spitting out the dose within the first minute of IP administration; or, vomiting within 30 minutes of IP administration | Up to 21 days of age
  Indicator of immediate post-ingestion tolerability of the investigational product
Frequency of maternal report of vomiting, abdominal distension, and/or diarrhea (during the period of IP administration). | Up to 21 days of age
  Indicator of post-ingestion tolerability of the investigational product
Frequency of IP not administered completely on a given day after one or two attempts due to intolerance. | Up to 21 days of age
  Indicator of incomplete or failed dose administration due to intolerance
Frequency of maternal report of colic-type symptoms (fuss/crying) | Up to 21 days of age
  Indicator of post-ingestion tolerability of the investigational product
Anthropometric outcomes: Length for age z-scores (LAZ) | Up to 6 months of age
  Z-scores generated based on raw lengths and INTERGROWTH-21st or World Health Organization growth standards.
Anthropometric outcomes: Weight for age z-scores (WAZ) | Up to 6 months of age
  Z-scores generated based on raw weights and INTERGROWTH-21st or World Health Organization growth standards.
Anthropometric outcomes: Weight-for-length z-scores (WLZ) | Up to 6 months of age
  Z-scores generated based on raw lengths and weights and INTERGROWTH-21st or World Health Organization growth standards.
Anthropometric outcomes: Head circumference for age z-scores (HCAZ) | Up to 6 months of age
  Z-scores generated based on raw head circumferences and INTERGROWTH-21st or World Health Organization growth standards.
Incidence of severe infection | Up to 60 days of age
  "Severe infection" (clinical outcome) defined as: at least one sign of clinical severe infection (CSI) (i.e., poor feeding, lethargy, convulsions, severe chest in-drawing, fever, or hypothermia) documented by a physician and/or physician diagnosis of sepsis or another serious bacterial infection (SBI); and at least one of the following two criteria: 1) physician decision to admit to hospital, administration of at least one dose of a parenteral antibiotic on the day when CSI/sepsis/SBI is first ascertained, and treatment with parenteral antibiotics for at least 5 days or 2) blood and/or cerebrospinal fluid culture positive for a pathogenic bacterial or fungal organism
Other clinical outcomes: Non-injury death | Up to 6 months of age
  Death due to any cause except death that was directly caused by physical trauma (medically certified cause of death and/or verbal autopsy) based on mother/caregiver report
Other clinical outcomes: Acute diarrhea | Up to 6 months of age
  Maternal/caregiver report of ≥3 loose stools in 24 hours for <14 days, using the modified Amsterdam scale
Other clinical outcomes: Persistent diarrhea | Up to 6 months of age
  Maternal/caregiver report of frequency and consistency of stool (≥3 loose stools in 24 hours for ≥14 days) using the modified Amsterdam scale
Other clinical outcomes: Vomiting | Up to 6 months of age
  Any vomiting as reported by mother/caregiver
Other clinical outcomes: Persistent vomiting | Up to 6 months of age
  Vomiting ≥3 times in a 24 hour period as reported by mother/caregiver.
Other clinical outcomes: Hospitalization | Up to 6 months of age
  Any inpatient admission for acute illness; excludes admission for elective surgical procedures
Other clinical outcomes: Cry/fuss | Up to 6 months of age
  Cry/fuss pattern questionnaire (up to 3-months of age) based on mother/caregiver report
Iron status and antioxidant capacity-related biomarkers: Stool | Up to 3 months of age
  Total iron in stool samples at day 14 of life (µg of iron/g dry weight of feces) as measured by atomic absorption spectrometry
Iron status-related biomarkers: Blood | Up to 3 months of age
  Serum ferritin (µg/L). Other measures if feasible: soluble transferrin receptor (mg/L) and hepcidin (ng/ml) at day 60 of age (approx.)
Average absolute and relative stool abundance (as defined above) of L. plantarum ATCC 202195 detected in non-supplemented siblings and mothers of infants who received the IP. | Up to 60 days of life (of enrolled infant)
  Indicator of environmental contamination by investigational product
Average number of intended doses received, irrespective of timing of dose | Up to 21 days of age
  Indicator of adherence to investigational product
Average proportion of doses received by day 10 of life | Up to 10 days of age
  Indicator of adherence to investigational product
Average proportion of doses received on scheduled day | Up to 21 days of age
  Indicator of adherence to investigational product
Average range (in days) between first and last dose | Up to 21 days of age
  Indicator of adherence to investigational product
Frequency of participant loss to follow-up | Up to 9 months of age
  Indicator of success of participant follow-up. Loss to follow-up defined as: 1) study personnel conclusively determine that a participant cannot be further contacted for the purposes of data collection for the remaining duration of scheduled follow-up visits OR 2) three months have passed since the scheduled but missed 6-month postnatal visit.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roth, MD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Bangladesh (2):
  - Maternal Child Health Training Institute, Dhaka
  - Mohammadpur Fertility Services Training Centre, Dhaka

IPD SHARING:
Plan to Share IPD: Yes
A detailed data sharing plan will be developed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: To be determined
Access Criteria: To be determined.

REFERENCES:
- [Derived] Pell LG, Qamar H, Bassani DG, Heasley C, Funk C, Chen C-Y, Shawon J, O'Callaghan KM, Pullenayegum E, Hamer DH, Haque R, Kabir M, Ahmed T, O'Kelly C, Hossain MI, Khan AZ, Loutet MG, Islam MS, Morris SK, Shah PS, Sherman PM, Sultana S, Mahmud AA, Saha SK, Sarker SA, Roth DE. Neonatal administration of Lactiplantibacillus plantarum ATCC 202195 with or without fructooligosaccharide in Bangladesh: a placebo-controlled randomized trial. mSphere. 2025 Mar 25;10(3):e0103224. doi: 10.1128/msphere.01032-24. Epub 2025 Feb 24. PMID 39992135